CLINICAL TRIAL: NCT04262765
Title: Open Label, Comparative, Multiple-dose, Fixed-sequence Steady State Trial in Healthy Volunteers to Assess the Pharmacokinetic Interaction of Ramipril, Atorvastatin and Amlodipine After a Multiple Oral Dose Administration
Brief Title: Drug-drug-interaction Study of Ramipril, Amlodipine and Atorvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Midas Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAAMAT-T1018/66
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
Keywords: ramiprilat; ramipril; amlodipine; atorvastatin; drug interaction; multiple-dose; pharmacokinetic
MeSH Terms: interventions — Ramipril; Amlodipine; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Subjects are to be admitted the night before dose no. 1 administration, confining at clinical site until the 24 hours post dose no. 5 administration. 4-days off interval between last dose of treatment A and first dose of treatment B allowed. Subjects to be admitted the night before dose no. 6 administration, confining at clinical site until the 24 hours post dose no. 10 administration. 4-days off interval between last dose of treatment B and first dose of treatment C allowed. Subjects to be admitted the night before dose no. 11 administration, confining at clinical site until the 24 hours post dose no. 26 administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment A-B-C-ABC (Experimental): The demographic characteristics of the 18 male subjects were as follows:
  * Age: 18-49 years
  * Weight: 55-105 kg
  * Height: 163-188 cm
  * BMI 18.5-29.9 kg/m²
  Interventions: Drug: Ramipril, Amlodipine and Atorvastatin

INTERVENTIONS:
Drug: Ramipril, Amlodipine and Atorvastatin — compare the pharmacokinetic of ramipril (and ramiprilat), atorvastatin as atorvastatin calcium trihydrate, amlodipine as amlodipine besilate from reference products given as a multiple dose

SUMMARY:
Study to determine the potential pharmacokinetic interaction of ramipril (and ramiprilat), atorvastatin as atorvastatin calcium trihydrate and amlodipine as amlodipine besilate at steady state after a multiple oral administration and to monitor the safety of the co-administration of these drugs. This study aims to determine if the steady state study pharmacokinetic parameters of any of the given drugs and the tolerability is altered when administered concomitantly.

DETAILED DESCRIPTION:
This study was an open-label, comparative, multiple-dose, fixed sequence steady state trial to compare the pharmacokinetic of ramipril, atorvastatin as atorvastatin calcium trihydrate, amlodipine as amlodipine besilate given as a multiple dose under fasting conditions in the absence and presence of each other.

Bioanalysis of ramipril, ramiprilat, atorvastatin and amlodipine is performed by LC/MS/MS method.

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasian, aged 18 to 50 years, inclusive.
* Body Mass Index (BMI) range within 18.5 - 30.0 Kg/m2.
* Physically and mentally healthy as judged by means of medical and standard laboratory examinations. Medical demographics performed not longer than two weeks before the initiation of the clinical study with significant deviations from the normal ranges.
* Standard ECG assessment is normal
* Informed consent given in written form according to chapter 5.3 of the study protocol.

Exclusion Criteria:

* Known allergy to the drugs under investigation or any ingredients or any other related drugs.
* Participation in a relative bioavailability study or in a clinical study within the last 80 days before first study drug administration or blood donation
* Presence of any clinically significant results from laboratory tests, vital sign assessment and electrocardiogram as judged by the investigator. Laboratory tests are performed not longer than two weeks before the initiation of the clinical study.
* Results of CPK or liver or kidney function tests which are outside the reference range.
* Hb test lower than 13.3 g/dl.
* Positive serologic findings
* History of drug or alcohol abuse.
* Subject is a heavy smoker.
* Subject has a history of significant asthma, peptic or gastric ulcer, sinusitis, pharyngitis, renal disorder (impaired renal function), hepatic disorder (impaired hepatic function), cardiovascular disorder, neurological disease such as epilepsy, haematological disorders or diabetes, psychiatric, dermatologic or immunological disorders.
* Subject having at screening examination a sitting blood pressure of less than 110/70 mm Hg or more than or equal to 140/90 mm Hg.
* Subjects who are known or suspected: not to comply with the study directives, not to be reliable or trustworthy, not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed, to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the unpleasantness they may be involved in.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-23 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration at steady state | up to 24 hours post-administration at steady state
  Maximum plasma concentration, it is read directly from the raw data
Area under the Plasma concentration curve (AUC0-t) | up to 24 hours post-administration at steady state
  Area under the plasma concentration curve from time 0 to the last measured (AUC0-t)

SECONDARY OUTCOMES:
Safety measurement (Adverse Events) | complete study, Day 1 until Day 31 (Follow-up)
  All observed or volunteered safety events regardless of treatment group or suspected causal relationship to the investigational product(s) will be reported during study.
Time until Cmaxss is reached (tmaxss) | up to 24 hours post-administration at steady state
  Time until Cmax is reached, it is read directly from the observed concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Bader, Study Director — International Pharmaceutical Research Center, Jordan
Locations (1):
- International Pharmaceutical Research Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No